CLINICAL TRIAL: NCT00926185
Title: A Phase 2, Multicenter, Randomized, Double-Masked and Placebo-Controlled Study Evaluating the Efficacy of Three Different Concentrations (0.1%, 1.0%, 5.0%) of SAR 1118 Ophthalmic Solution in Subjects With Dry Eye Using the Controlled Adverse Environment (CAE) Model
Brief Title: A Study Evaluating the Efficacy of SAR 1118 (0.1%, 1.0%, 5.0%) Ophthalmic Solution in Subjects With Dry Eye Conducted in a Controlled Adverse Environment (CAE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1118-KCS-100
Record Dates: First submitted 2009-06-20; First posted 2009-06-23 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Dry Eye
Keywords: Dry Eye; ophthalmic delivery
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo Ophthalmic Solution
  Interventions: Drug: Placebo
- 0.1% Lifitegrast (Experimental): Lifitegrast
  Interventions: Drug: Lifitegrast
- 1.0% Lifitegrast (Experimental): Lifitegrast
  Interventions: Drug: Lifitegrast
- 5.0% Lifitegrast (Experimental): Lifitegrast
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Lifitegrast — Ophthalmic Solution
  Other Names: SAR 1118
  Arms: 0.1% Lifitegrast; 1.0% Lifitegrast; 5.0% Lifitegrast
Drug: Placebo — Ophthalmic Solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of three different concentrations (0.1%, 1.0%, 5.0%) of SAR 1118 Ophthalmic Solution compared to placebo in the treatment of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form and HIPAA document
* Willing and able to comply with all study procedures
* Be at least 18 years of age
* Patient-reported history of dry eye in both eyes
* Demonstrate a positive response when exposed to the Controlled Adverse Environment model
* A negative urine pregnancy test if female of childbearing potential and must use adequate birth control throughout the study period

Exclusion Criteria:

* Any ocular condition that, in the opinion of the Investigator, could affect study parameters including, but not limited to, active ocular infection, ocular inflammation, glaucoma, and/or diabetic retinopathy
* Unwilling to avoid wearing contact lenses for 7 days prior to and for duration of the study period
* Any blood donation or significant loss of blood within 56 days of Visit 1
* Any history of immunodeficiency disorder, positive HIV, hepatitis B, C, or evidence of acute active hepatitis A (anti-HAV IgM), or organ or bone marrow transplant.
* Use of any topical ophthalmic preparations (including tear substitutes) 72 hrs prior to screening assessments and through the entire study period
* Any significant illness that could interfere with study parameters
* History of laser-assisted in situ keratomileusis (LASIK) or similar type of corneal refractive surgery within 12 months prior to Visit 1, and/or any other ocular surgical procedure within 12 months prior to Visit 1; or any scheduled ocular surgical procedure during the study period.
* Known history of alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2009-08-03 (Actual); Primary Completion 2010-02-18 (Actual); Study Completion 2010-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - The Eye Care Group, Waterbury, Connecticut
  - Central Maine Eye Care, Lewiston, Maine
  - Ora, Inc. (two locations), Andover, Massachusetts
  - Mundorf Eye Center, Charlotte, North Carolina
  - Total Eye Care, P.A., Memphis, Tennessee

REFERENCES:
- [Derived] Semba CP, Torkildsen GL, Lonsdale JD, McLaurin EB, Geffin JA, Mundorf TK, Kennedy KS, Ousler GW. A phase 2 randomized, double-masked, placebo-controlled study of a novel integrin antagonist (SAR 1118) for the treatment of dry eye. Am J Ophthalmol. 2012 Jun;153(6):1050-60.e1. doi: 10.1016/j.ajo.2011.11.003. Epub 2012 Feb 11. PMID 22330307

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in a Controlled Adverse Environment (CAE).
Period: Overall Study
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Started | 57 | 57 | 58 | 58
Completed | 54 | 51 | 48 | 48
Not Completed | 3 | 6 | 10 | 10

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo | Total
Number analyzed (Participants) | 57 | 57 | 58 | 58 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.14 (13.100) | 63.63 (11.883) | 62.26 (12.220) | 60.38 (12.930) | 62.34 (12.523)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 40 | 47 | 45 | 179
  Male | 10 | 17 | 11 | 13 | 51

OUTCOME MEASURES:

1. Primary Outcome: Inferior Corneal Fluorescein Staining Score in Pre-Controlled Adverse Environment at Day 84
Description: Corneal staining was performed to grade the degree of corneal epithelial cell injury as measured by fluorescence using slit-lamp examination. The staining was graded with the Ophthalmic Research Associates, Inc. (ORA) scale. The corneal surface is divided into three regions: superior, central and inferior. The scores for each of these 3 regions ranged from 0 to 4 (0=no staining; 1=occasional; 2=countable; 3=uncountable, but not confluent; 4=confluent) with 0.5 point increments, and lower score indicates a better outcome. Inferior corneal fluorescein staining scores from the study eye only were reported. Study eye is the 'worse eye', defined as the eye with worse (higher) score at baseline.
Time Frame: Day 84
Population: Intent-to-treat (ITT) population with LOCF defined as all randomized subjects. For the efficacy analysis, the Last Observation Carried Forward (LOCF) method will be used to impute missing values.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 57 | 55 | 54 | 55
units on a scale | 2.03 (0.868) | 1.92 (0.768) | 1.83 (0.680) | 2.05 (0.715)
Statistical Analysis 1: Comparison: Lifitegrast 0.1% vs Placebo; Test type: Superiority or Other; p = 0.9381, Dunnett's test; Treatment Effect = 0.06, 95% CI 2-sided [-0.26 to 0.39] — Analysis of covariance model with treatment, baseline, and site
Statistical Analysis 2: Comparison: Lifitegrast 1.0% vs Placebo; Test type: Superiority or Other; p = 0.3585, Dunnett's test; Treatment Effect = 0.20, 95% CI 2-sided [-0.13 to 0.53] — Analysis of covariance model with treatment, baseline, and site
Statistical Analysis 3: Comparison: Lifitegrast 5.0% vs Placebo; Test type: Superiority or Other; p = 0.1375, Dunnett's test; Treatment Effect = 0.27, 95% CI 2-sided [-0.06 to 0.60] — Analysis of covariance model with treatment, baseline, and site

2. Secondary Outcome: Inferior Corneal Staining Score Change From Baseline (CFB) to Day 84
Description: as for outcome 1
Time Frame: Baseline (Day 0) and Day 84
Population: ITT set with LOCF was used for analysis of this outcome. Here, "n" signifies the number of participants evaluable for the respective time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Number analyzed (Participants) | 57 | 57 | 58 | 58
units on a scale
  Pre-CAE: Baseline: number analyzed (Participants) | 57 | 56 | 58 | 58
  Pre-CAE: Baseline | 1.78 (0.473) | 1.82 (0.508) | 1.77 (0.515) | 1.65 (0.513)
  Pre-CAE: CFB to Day 84: number analyzed (Participants) | 57 | 55 | 54 | 55
  Pre-CAE: CFB to Day 84 | 0.25 (0.841) | 0.10 (0.735) | 0.05 (0.773) | 0.40 (0.802)
  Post-CAE: Baseline: number analyzed (Participants) | 57 | 56 | 58 | 58
  Post-CAE: Baseline | 3.18 (0.417) | 3.28 (0.610) | 3.16 (0.523) | 3.04 (0.602)
  Post-CAE: Day 84: number analyzed (Participants) | 57 | 55 | 54 | 55
  Post-CAE: Day 84 | 2.86 (0.962) | 2.88 (0.860) | 2.90 (0.918) | 2.62 (0.855)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until the end of follow-up visit, up to Day 86
Arm/Group | Lifitegrast 0.1% | Lifitegrast 1.0% | Lifitegrast 5.0% | Placebo
Serious Adverse Events (participants affected / at risk) | 2/57 | 1/57 | 0/58 | 1/58
Other Adverse Events (participants affected / at risk) | 20/57 | 13/57 | 40/58 | 11/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast 0.1% (N=57) | Lifitegrast 1.0% (N=57) | Lifitegrast 5.0% (N=58) | Placebo (N=58)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifitegrast 0.1% (N=57) | Lifitegrast 1.0% (N=57) | Lifitegrast 5.0% (N=58) | Placebo (N=58)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Visual acuity reduced (Eye disorders) | 6 (7) | 2 (3) | 1 (1) | 3 (3)
Instillation site irritation (General disorders) | 7 (7) | 5 (5) | 20 (20) | 6 (6)
Instillation site pain (General disorders) | 6 (6) | 3 (3) | 20 (20) | 3 (3)
Instillation site reaction (General disorders) | 0 (0) | 1 (2) | 8 (16) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (3) | 7 (12) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicentre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicentre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.